CLINICAL TRIAL: NCT05023798
Title: Development Study to Undertake a Comprehensive Performance Evaluation of Prototype Non-Invasive Blood Glucose Measurement Systems Compared to a Standard (Invasive) Measurement Method of Blood Glucose
Brief Title: Study to Evaluate a Prototype Non-Invasive BG Measurement System
Acronym: ATD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Afon Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: 04-001
Record Dates: First submitted 2021-08-09; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: diabetes; non-invasive; BG sensor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- ATD Cohort 1: The first iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment.
  Interventions: Device: ATD (device test)
- ATD Cohort 2: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 3: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 4: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 5: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 6: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 7: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 8: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 9: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)
- ATD Cohort 10: The next iteration of the sensor will be tested and results compared to the gold-standard laboratory measuring equipment. The prototype will be tested on a cohort of 3-5 patients.
  Interventions: Device: ATD (device test)

INTERVENTIONS:
Device: ATD (device test) — Medical device test (no intervention)

SUMMARY:
1. Diabetes mellitus is a chronic disease currently affecting more than 425 million people, of which one-third are people older than 65 years. In the UK, the number of people currently diagnosed with diabetes surpassed 3.8 million in 2019, with someone being diagnosed with the illness every two minutes (Diabetes.org figures). The prototype device being tested is a non-invasive blood glucose measurement system worn on the wrist. This would help people with diabetes manage their condition better and help prevent complications.
2. The main objectives of the research are:

   1. To determine how accurate and effective the Afon prototype non-invasive blood glucose measurement system is, as compared to a gold standard invasive method.
   2. To chart the Afon device's predicted blood glucose levels over time.
3. The study will be done with 30-50 patients. Eligible patients will have been diagnosed with diabetes (type 1 or 2) at least one year prior, be between 18 and 80 years old, and with a BMI between 18-35 kg/m2. For details of the full list of inclusion and exclusion criteria, see accompanying documentation.
4. The trial will be conducted at the Joint Clinical Research Facility (JCRF), Institute of Life Science 2, Swansea University, SA2 8PP.
5. Participants will attend the site for a total of 5 visits, one for screening, and four study visits, no more than 7 days apart. The study will run for one year.

DETAILED DESCRIPTION:
Diabetes is a chronic disease currently affecting more than 425 million people worldwide. In the UK, the number of people currently diagnosed with diabetes surpassed 3.8 million in 2019, with someone being diagnosed with the illness every two minutes (Diabetes.org figures).By the end of this year, 4 million deaths will happen worldwide as a result of diabetes and its complications. These complications include renal failure, blindness, and amputation. It is well established clinically that good glycaemic control minimises the risk of long-term complications and improves morbidity and mortality. Current problems with frequent blood glucose testing are mainly due to patient intolerability. Many patients find finger prick testing for blood glucose levels to be painful, dislike using sharp objects and seeing their own blood. There is also a risk of infection, and in the long term, this practice can result in damage to the finger tissue. This is because the fingers have a high concentration of sensory nerve endings. Additionally, the current invasive blood glucose monitoring systems suffer limitations in terms of the requirement for continuous calibration and susceptibility to contamination by the growth of various living organisms.

The Afon technology device would be a gamechanger in terms of improving the quality of life of millions of patients and improve their chances to manage the condition without severe complications.

ELIGIBILITY:
Inclusion Criteria:

Patient who has a documented Type 1 diagnosis (diagnosed under age 29), or Type 2 diabetes for more than one year (with negative GAD antibody test results) and who are willing and able to give informed consent for participation in the study Male or female patient Patient aged 18 to 80 years Patients with a BMI 18-35 kg/m2.

Exclusion Criteria:

The patient may not enter the study if ANY of the following apply:

Type 1 patients diagnosed after age 29 Type 2 patients with positive GAD antibody test results Patient with other active implantable medical devices, such as pacemakers Patient who is currently participating in another clinical trial for a pharmaceutical product Patient with a history of allergy to any materials used in the prototype sensors or materials used to stabilise the devices or cabling including Rocktape, double-sided tape and prosthetic adhesive Female patient who is pregnant or lactating

* Patient with any injury or infection of the wrist
* Patient who is unwilling or unable to attend each visit fasting from midnight (water is permitted freely) or fasting for a minimum of 3 hours (for an afternoon session)
* Patient who takes paracetamol or aspirin in the 24 hours preceding each visit
* Patient with clinically significant abnormal values in clinical chemistry, as judged by the PI
* Concurrent illness or a condition that may interfere with blood glucose levels (e. g. carcinoma, haematological disease, vasculitis, connective tissue disease, alcohol neuropathy)
* Patient who is incapable of giving informed legal consent
* Recent (1 month) episode of DKA, HONK or severe hypoglycaemia
* Patient on pramlintide (Symlin/Tripro-Amylin)
* Patient who attends the visit under the influence of alcohol or recreational drugs
* Patient with severe macrovascular disease - stroke, CVD, CKD stage IV -V Patient who fails screening for alcohol and recreational drugs use.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Trial participants will be patients who have agreed to help with the development of a non-invasive glucometer. Between thirty and fifty patients will be enrolled in this pilot study of prototype sensors. If any prototype sensor is of interest and promise, the number of patients exposed to it may be increased. Subjects who withdraw from the study will be replaced.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Exploratory Efficacy Objective 1 | Up to 4 hours per test session.
  To estimate real-time serial blood glucose levels from the device measurements using a gold standard methodology for blood glucose measurement as control.
  A comparison addressing the potential differences of MARDs and PARDs respectively will be done for the Afon system tested and assessed using mixed effect linear models with the BG as the fixed effect and subjects as random effects. Within the model the least square means, the differences between least square means of MARD of the Afon system and corresponding two-sided 95% parametric confidence interval will be calculated.
Exploratory Efficacy Objective 2 | Up to 4 hours per test session.
  To chart patient-specific predicted vs actual blood glucose levels over time, including before and after glucose challenge.
  The type I error is set at 5% two-sided.
Safety Objective 1 | Up to 4 hours per test session.
  To examine the safety and tolerability of the prototype sensors.
  Number of participants with no device-related SAE = 0.
Exploratory Usability Objective | 25 minutes - 1 hour during a test session.
  To obtain patient input for wearable device design by means of a usability questionnaire1 answered questionnaire per participant.

CONTACTS AND LOCATIONS:
Locations (1):
- JCRF, Swansea, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data will be shared.

REFERENCES:
- [Derived] Handy C, Chaudhry MS, Qureshi MRA, Love B, Shillingford J, Plum-Morschel L, Zijlstra E. Noninvasive Continuous Glucose Monitoring With a Novel Wearable Dial Resonating Sensor: A Clinical Proof-of-Concept Study. J Diabetes Sci Technol. 2024 Nov;18(6):1408-1415. doi: 10.1177/19322968231170242. Epub 2023 Apr 27. PMID 37102600